CLINICAL TRIAL: NCT03082352
Title: Clinical Bioequivalence Study on Two Metoprolol Tablet 100mg Formulations
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bright Future Pharmaceuticals Factory O/B Bright Future Pharmaceutical Laboratories Limited (Industry)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BABE-P15-100
Record Dates: First submitted 2017-03-12; First posted 2017-03-17 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Healthy
MeSH Terms: interventions — Metoprolol

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BF-Metoprolol Tablet 100mg (Experimental): During the study session, healthy subjects will be administered a single dose of BF-Metoprolol Tablet 100mg after an overnight fast of approximately 10 hours
  Interventions: Drug: BF-Metoprolol Tablet 100mg
- Betaloc Tablet 100mg (Active Comparator): During the study session, healthy subjects will be administered a single dose of Betaloc Tablet 100mg after an overnight fast of approximately 10 hours
  Interventions: Drug: Betaloc Tablet 100mg

INTERVENTIONS:
Drug: BF-Metoprolol Tablet 100mg — BF-Metoprolol Tablet 100mg is a generic product manufactured by Bright Future Pharmaceuticals Factory O/B Bright Future Pharmaceutical Laboratories Limited
  Other Names: Metoprolol Tablet 100mg
  Arms: BF-Metoprolol Tablet 100mg
Drug: Betaloc Tablet 100mg — Betaloc Tablet 100mg will be used as a comparator drug for the BE study
  Other Names: Metoprolol Tablet 100mg
  Arms: Betaloc Tablet 100mg

SUMMARY:
The purpose of the study is to compare the bioavailability of a generic product of metoprolol with that of a reference product when administered to healthy volunteers under fasting conditions. The test product is BF-Metoprolol Tablets 100mg manufactured by Bright Future Pharmaceuticals Factory O/B Bright Future Pharmaceutical Laboratories Limited and the reference product is Betaloc Tablet 100mg. The plasma kinetic data of metoprolol obtained from two formulations will be used to access the interchangeability of the products.

DETAILED DESCRIPTION:
The study design is a single-dose, two-treatment, two-period, two-sequence cross over with a washout period of one to two weeks. Subject will be randomly assigned to two groups corresponding to two dosing sequences. Each subject will undergo two study (treatment) sessions, during which a single oral dose of 100mg metoprolol from either test or reference formulations will be administered. The estimated duration of subject's participation will be about 29-36 days (i.e. 3 weeks for screening and medication restraint, 1 day each for study (treatment) sessions I and II, 1 - 2 weeks as washout period. Venous blood samples will be collected at pre-dose (0h), and up to 24h post dose. The plasma concentrations of metoprolol will be determined by a validated assay. The non-compartmental method will be used to analyze the plasma concentration-time data and calculate the main pharmacokinetic parameters such as Cmax, Tmax, AUC0-last, AUC0-inf, and T1/2. ANOVA will be calculated on logarithmically transformed Cmax, AUC0-last and AUC0-inf. The two one sided tests will be used to calculate the 90% confidence intervals for the mean difference in AUC0-last, AUC0-inf and Cmax and to assess the bioequivalence of the two products

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female, 18 to 55 years of age
* Body Mass Index between 18 to 30 kg/m2
* Accessible vein for blood sampling
* High probability for compliance and completion of the study
* Female subjects must agree to practice abstinence or take effective contraceptive methods to prevent pregnancy from the start of the screening and until two weeks of last dose administration

Exclusion Criteria:

* Clinically significant hepatic, renal, biliary, cardiovascular, gastrointestinal, haematological and other chronic and acute diseases within 3 months prior to the study
* Clinically significant abnormality in physical examination, vital sign, laboratory test results, ECG evaluation, urine test, blood chemistry or haematological test
* Regular consumption of tobacco used in any forms
* Regular consumer of alcohol (more than one drink per day)
* Blood donation within 4 weeks prior to the start of the study
* Use of metoprolol within 4 weeks before the study
* Use of antihypertensive medications or other beta blockers within 4 weeks before the study
* Volunteer in any other clinical drug study within 2 months prior to this study
* Hypersensitivity to metoprolol or other drugs in its class
* History of drug abuse in any form
* Female subjects who are breastfeeding or pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of metoprolol | 24 hours
Area under the plasma concentration versus time curve (AUC) of metoprolol | 24 hours

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) of metoprolol | 24 hours
Elimination half-life (t1/2) of metoprolol | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Zuo, Principal Investigator — School of Pharmacy, The Chinese University of Hong Kong; Riza Ozaki, Study Director — Phase 1 Clinical Trial Centre, The Chinese University of Hong Kong; Brian Tomlinsion, Study Director — Department of Medicine and Therapeutics, The Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Study investigators and his/her study team members, domestic and foreign regulatory agencies, the IRB/EC involved in the study, and laboratories and other individuals and organizations that analyze the subjects' protected health information in connection with this study have access to the data or study